CLINICAL TRIAL: NCT01262040
Title: Narrow Band Imaging (NBI): A Novel Imaging Modality in Minimally Invasive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-180
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cancer; Gastrointestinal Carcinoma; Pancreatic Carcinoma; Lung Cancer; Esophageal Carcinoma
Keywords: NBI; ENDOMETRIUM; FALLOPIAN TUBE; OVARY; PERITONEUM; Surgery; Lung; Pancreatic; Esophageal; thorascopic; laparoscopic; robotic; 10-180
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Esophageal Neoplasms | interventions — Narrow Band Imaging

ARMS (1):
- pts having a thorascopic, laparoscopic or robotic procedure (Experimental): The procedure will begin with washings (peritoneal) and two assessments of the extent of peritoneal disease. First, a four quadrant inspection of the peritoneal cavity under white light, this is the standard of care assessment. Then, a repeat four quadrant inspection of the peritoneal cavity under NBI will be done, this is the only experimental component of the design. White light imaging will always be done first, followed by NBI. For those patients scheduled for thorascopic procedures: The procedure will begin with sampling of pleural effusions when clinically indicated. Then there will be two assessments of the pleural surfaces. First, an inspection of the pleural cavity under white light, this is the standard of care assessment. Then, a repeat inspection under NBI, this is the only experimental component of the design. White light imaging will always be done first, followed by NBI.
  Interventions: Other: Narrow Band Imaging (NBI)

INTERVENTIONS:
Other: Narrow Band Imaging (NBI) — The intervention is visual assessment of the peritoneal or pleural surface with NBI followed by biopsy and photographic documentation of any abnormal lesions. Photograph or video of abnormality(ies) under white light and NBI.

SUMMARY:
The purpose of this study is to determine whether narrowband imaging (NBI) makes it easier for a surgeon to see cancer.

NBI is a kind of light. Normally, white light is used during surgery. White light uses many wavelengths of light. NBI only uses two wavelengths which highlight the blood vessels. This makes it easier for the surgeon to see blood vessels. Tumors often have more blood vessels than normal tissue. As a result, NBI may make it easier for the surgeon to see small tumors.

In this study the surgeon will look with both normal white light and NBI. This way a comparison can be made to determine which is superior.

Improved identification of tumors allows doctors and patients to make informed decisions about whether treatment is needed after surgery. It also provides additional information to determine which treatments may be best.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet one (or more) of the following criteria:
* Preoperative diagnosis of ovarian, fallopian tube, or primary peritoneal carcinoma (all stage, grade and histology)
* Preoperative diagnosis of grade III endometrial carcinoma (all stage, all histology)
* Preoperative diagnosis of uterine serous carcinoma (all stage, all grade)
* Preoperative diagnosis of clear cell endometrial carcinoma (all stage, all grade)
* Preoperative diagnosis of endometrial carcinosarcoma (all stage, all grade)
* Gastrointestinal carcinoma (all histology, stage and grade)
* Pancreatic carcinoma (all histology, stage and grade)
* Lung cancer (all histology, stage and grade)
* Esophageal carcinoma (all histology, stage and grade)
* Suspected or pathologically confirmed metastatic disease to the lung (all disease primaries)
* Suspected or pathologically confirmed malignant pleural effusion (all disease primaries)

Patients must meet all of the following criteria:

* Planned thorascopic robotic or laparoscopic surgical approach
* >18 years old
* Not pregnant
* Able to give consent Participation in other research protocols does not exclude a patient from participation in this study.

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-12-14 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of Narrow Band Imaging (NBI) at the time of thorascopic, laparoscopic or robotic surgery. | 1 year

SECONDARY OUTCOMES:
Determine what percentage of patients have surface metastasis identified with NBI that were not seen on white light imaging. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Abu-Rustum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm